CLINICAL TRIAL: NCT04813328
Title: A Pilot Study of the Effects of Helminth Infection and SARS-CoV-2 Seropositivity on Immune Response and the Intestinal Microbiota in India
Brief Title: The Effect of Helminth Infection Plus COVID-19 Infection on the Immune Response and Intestinal Microorganisms
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: SARS-CoV-2/helminth
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Coded PBMC, serum, stool RNA samples and data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot, cross-sectional, sample collection study to characterize the immune response and intestinal microorganisms in people with and without COVID-19 antibodies and helminth infection.

DETAILED DESCRIPTION:
This is a pilot, cross-sectional, sample collection study to characterize the immune response and intestinal microbiota in people with and without SARS-CoV-1 antibodies and helminth infection.

A target sample size of 1500 participants aged 5 years or older will undergo a one-time blood and stool collection for SARS-CoV-2 antibody testing, diagnosis of parasitic infections, and experimental studies including transcriptomics (RNA) and microbiome (intestinal microorganisms) characterization. Participants willing to take part in the study will be selected from households in the Tiruvallur district, Tamil Nadu, India. Individual study participation involves a single study visit. Participants will be informed of the results of clinical testing and will be referred for medical care as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.

Exclusion Criteria:

* Poor venous access precluding venipuncture.
* History of any illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the participant's participation in the protocol, or compromise the scientific objectives.

Participants may be co-enrolled in other studies; however study staff should be notified of co-enrollment.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants will be enrolled from households in the Tiruvallur district, Tamil Nadu, India. Villages and towns in the Tiruvallur district will be selected in consultation with the Department of Public Health, Tamil Nadu. Areas that are known hotspots for COVID-19 will be selected.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with helminth infections | Day 1
  Measured by qPCR diagnostics of stool DNA extraction
Number of participants with SARS-CoV-2 antibodies | Day 1
  Measured by real-time qPCR (quantitative polymerase chain reaction) assay
Number of participants with positive malaria test | Day 1
  Measured by fingerprick blood samples
Average Differential blood count | Day 1
  Measured from venipuncture blood samples
Average Hematocrit levels | Day 1
  Measured from venipuncture blood samples
Number of participants with latent tuberculosis infection | Day 1
  Measured by IFN-γ release assay
Number of participants with Wuchereria bancrofti infection | Day 1
  Measured by enzyme-linked immunosorbent assay (ELISA)
Number of participants with Strongyloides stercoralis infection | Day 1
  Measured by enzyme-linked immunosorbent assay (ELISA)
Number of participants with Ascaris infection | Day 1
  Stool sample analysis DNA extraction for qPCR and 16S sequencing
Number of participants with hookworm infection | Day 1
  Stool sample analysis DNA extraction for qPCR and 16S sequencing
Number of participants with Strongyloides infection | Day 1
  Stool sample analysis using Baermann technique, DNA extraction for qPCR and 16S sequencing
Number of participants with Trichuris infection | Day 1
  Stool sample analysis using DNA extraction for qPCR and 16S sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Subash Babu, MBBS, PhD, Principal Investigator — National Institute for Research in Tuberculosis; P'ng Loke, PhD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institute for Research in Tuberculosis - International Centers for Excellence in Research (NIRT-ICER), Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Ferris BF, Balasubramanian S, Rajamanickam A, Munisankar S, Dasan B, Menon PA, Loke P, Babu S, Chami GF. Relative contribution of biomedical, demographic, and socioeconomic factors to COVID-19 vaccine receipt in rural India. PLoS One. 2024 Jun 24;19(6):e0305819. doi: 10.1371/journal.pone.0305819. eCollection 2024. PMID 38913614